CLINICAL TRIAL: NCT00103883
Title: A Novel Method to Determine HIV Incidence Among Youth
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: ATN 022
Record Dates: First submitted 2005-02-15; First posted 2005-02-16 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-02

CONDITIONS: HIV Infection
Keywords: HIV; Detuned Assay; Enzyme Immunoassay (EIA); HIV Incidence; Laboratory assay; Sensitive/Less sensitive Assay; Acute Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Phenotypic and genotypic testing for antiretroviral drug (ART) resistance will be done on stored samples from all subjects who are identified as recently infected by the serum based DV S/LS reference method. An assay for viral replication fitness will also be done on these same samples. This testing will provide a recent assessment of prevalence of transmitted ART resistant HIV-1 in this population.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV Infected Teens -ATN Clinical Sites: HIV infected teens who are referred to or engaged in care at any of the 15 ATN clinical sites during the course of the study.
- HIV Positive - ATN Clinical Sites: Youth who test HIV positive at ATN-managed or ATN-affiliated HIV Counseling and Testing Sites (CTS) during the course of the study.
- HIV Positive - BCHD STD Clinic: Youth who test HIV positive at the BCHD STD Clinic during the course of the study.

SUMMARY:
Identifying young people with early HIV-1 infection is important for increasing linkage to care, for behavioral counseling, and for enrolling individuals into programs that can provide effective interventions to disease progression and improve outcome. This study will develop and evaluate a saliva-based sensitive/less sensitive (S/LS) assay for differentiating persons with recent HIV-1 infection (less than 133 days) from those with established HIV-1 infection.

DETAILED DESCRIPTION:
HIV infection incidence estimates are important, not only for determining specific populations where community HIV education sessions can have the most benefit or where changes in infection patterns are occurring, but also to target these populations for therapeutic interventions and measure their effect in the community. It is estimated that half of all new HIV infections in the United States occur in persons under the age of 25 each year, translating to approximately 20,000 new HIV-infected young people annually.

Incidence can be estimated by testing a cohort of individuals for antibody at two different time periods and observing the number of new infections, or by demonstrating the presence of HIV p24 or viral RNA in antibody-negative persons. Since these strategies are logistically difficult, expensive, and/or require significant laboratory infrastructure, new laboratory-based strategies were devised that can classify individuals as recently infected or with established infection. These serologic assays are known as "sensitive/less sensitive (S/LS) assays". They are based on either the concept of antibody titer or the concept of antibody avidity. There are several S/LS tests available but all of them are performed on serum collected via venipuncture. Based on several studies showing that obtaining saliva is a more desirable method of collection for adolescents receiving HIV testing, it is anticipated that the collection of saliva and its use for determining HIV incidence by S/LS methods among adolescents would be a valuable adjunct for population studies and for increasing compliance for testing and enrollment.

The aim of this study is to prove equivalence between the serum S/LS reference method (CDC validated serum S/LS Dilutional Vironostika (DV) from Organon Teknika) and the experimental method that uses an FDA approved saliva collection device (OraSure Technologies). Our rationale follows a syllogism, i.e., if the serum S/LS EIA (DV) is the best serologic method to determine incidence estimates and a saliva S/LS method is found to perform equivalently, then it follows that the saliva S/LS method can be used effectively to determine incidence. Therefore, our purpose is to show equivalence between the two assays. To address the issue of accuracy, further studies are planned to assess the saliva S/LS test against seroconversion panels where the exact time of acquisition of HIV infection is known.

This is a cross-sectional, laboratory-based study designed to develop and evaluate a saliva-based S/LS assay for differentiating individuals with recent HIV infection (less than 133 days) from those with established HIV infection. A total of 440 subjects will be recruited in the study. A serum and two saliva samples will be obtained from every subject. The first 40 patient samples will be used to develop and calibrate the saliva-based S/LS method. The remaining patient samples will be tested using the calibrated saliva based S/LS assay and the reference serum S/LS assay and concordance between the two methods will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 through 24 years
* HIV infection determined by routine HIV testing strategies
* Ability to give informed consent or assent with parental permission, where required

Exclusion Criteria:

* Visibly distraught or emotionally unstable
* Intoxicated or under the influence of psychoactive agents
* First disclosure of sexual, physical, or emotional abuse
* Clinically presents as acutely ill

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Two hundred fifty subjects will be recruited from the fifteen sites of the Adolescent Trials Network for HIV/AIDS Interventions (ATN) and 190 from the BCHD STD Clinic, a sexually transmitted disease clinic of the Baltimore City Health Department (BCHD). The age range for subjects from the ATN clinical sites will be 12 through 24 years and those from the BCHD STD Clinic will be 17 through 30 years.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2003-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Phase I - Serum-based S/LS assay result | 15-20 Months
  To develop and calibrate a saliva S/LS assay using the FDA licensed OraSure collection device in conjunction with its matched saliva EIA assay to differentiate persons with recent versus established HIV infection (Phase I)
Phase II - Saliva-based S/LS assay result | 15-20 Months
  To assess that the saliva S/LS method performs equivalently to the reference serum S/LS method for HIV incidence estimates in populations of youth (Phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Ligia Peralta, MD, Study Chair — University of Maryland
Locations (15):
- United States (14):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - University of Maryland Medical School, Baltimore, Maryland
  - Childrens Hospital Boston, Boston, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- University Pediatric Hospital, San Juan, Puerto Rico